CLINICAL TRIAL: NCT02968498
Title: Blood Glucose Response After Oral Intake of Lactulose in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fresenius Kabi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Lact-001-CEN
Record Dates: First submitted 2016-11-16; First posted 2016-11-18 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Blood Glucose
Keywords: Blood glucose level; Oral intake; Lactulose; Healthy volunteers
MeSH Terms: interventions — Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study arm 1 (Active Comparator): Lactulose crystals 10 g vs lactulose crystals 20 g vs oral glucose 20 g vs still water
  Interventions: Dietary Supplement: Lactulose crystals 10 g; Dietary Supplement: Lactulose crystals 20 g; Dietary Supplement: Oral glucose 20 g; Dietary Supplement: Still water
- Study arm 2 (Active Comparator): Lactulose liquid 10 g vs lactulose liquid 20 g vs oral glucose 20 g vs still water
  Interventions: Dietary Supplement: Lactulose liquid 10 g; Dietary Supplement: Lactulose liquid 20 g; Dietary Supplement: Oral glucose 20 g; Dietary Supplement: Still water

INTERVENTIONS:
Dietary Supplement: Lactulose crystals 10 g — White or almost white crystalline powder used as food ingredient. The products will be provided in sachets to be dissolved in 250 mL water.
  Arms: Study arm 1
Dietary Supplement: Lactulose crystals 20 g — White or almost white crystalline powder used as food ingredient. The products will be provided in sachets to be dissolved in 250 mL water.
  Arms: Study arm 1
Dietary Supplement: Lactulose liquid 10 g — Clear, viscous liquid, colourless or pale brownish-yellow liquid syrup (solution). The products will be provided in sachets to be dissolved in 250 mL water.
  Arms: Study arm 2
Dietary Supplement: Lactulose liquid 20 g — Clear, viscous liquid, colourless or pale brownish-yellow liquid syrup (solution). The products will be provided in sachets to be dissolved in 250 mL water.
  Arms: Study arm 2
Dietary Supplement: Oral glucose 20 g — White crystalline powder used as food ingredient. To standardise for 20 g glucose, 22 g glucose monohydrate will be used. The products will be provided in sachets to be dissolved in 250 mL water.
  Other Names: glucose monohydrate
Dietary Supplement: Still water — Still water will be used. Water from the same source will be also used to dissolve investigational and control products.

SUMMARY:
Prospective, open, mono-center, randomized, two part study with 4-way cross-over design in each study part.

The objective of the study is to investigate blood glucose levels after oral intake of defined amounts of lactulose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Age: 18-65 years
* Approx. 3-5 bowel movements per week
* Caucasian
* Availability and presence in the trial unit for approx. 4 hours/ week for 4 times in a row with approx. 1 week of washout in between
* Signed informed consent form

Exclusion Criteria:

* Known (family) history of diabetes mellitus or use of anti-hyperglycaemic drugs or Insulin
* Clinically relevant renal or hepatic disease, liver enzymes > 10% above reference range
* Fasting blood glucose > 100 mg/dL or HbA1c outside of reference range
* Total cholesterol > 250 mg/dL or triglycerides > 150 mg/dL
* Haemoglobin < 11 g/dL (women); < 12.5 g/dL (men)
* BMI < 19 kg/m² and ≥ 30 kg/m²
* Intentional and unintentional weight loss > 5% in the previous 6 months
* Smoker
* Major medical or surgical event requiring hospitalization within the previous 3 months
* Presence of disease or drug(s) influencing digestion and absorption of nutrients or bowel habits
* Intake of medications known to affect glucose tolerance, e.g., steroids, protease inhibitors or antipsychotics (stable doses of e.g., oral contraceptives, thyroxin, vitamins and mineral supplements or drugs to treat hypertension or osteoporosis are acceptable)
* Chronic intake of substances affecting blood coagulation (e.g. acetylic acid, anticoagulants, diuretics, thiazides), which in the investigator's opinion would impact volunteer safety
* Hereditary problems of galactose or fructose intolerance, lactase deficiency or glucose-galactose malabsorption
* Suspicion of drug abuse
* Abuse of alcoholic drinks, defined as an average daily intake of more than one litre of beer per day or equivalent amount of alcohol in other beverages
* Pregnant or breast feeding women
* Known or suspected allergy to any component of the investigational product(s)
* Known HIV-infection
* Known acute or chronic hepatitis B and C infection
* Blood donation within 4 weeks prior to visit 1 or during the study
* Volunteer unable to co-operate adequately
* Participation in a clinical trial with an investigational product within one month before start of study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-11; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Capillary blood glucose levels as incremental area under the curve (iAUC) above baseline (iAUC(0-180min)) | 0-180 min

SECONDARY OUTCOMES:
Maximum blood glucose concentration (Cmax) | 0-180 min
Maximum increase of blood glucose concentration (Max_increase) | 0-180 min
  Cmax minus baseline value
Relative maximum increase of blood glucose concentration(Max_increase rel) | 0-180 min
  Cmax / baseline value
Time to reach maximum blood glucose concentration (Tmax) | 0-180 min
First time to reach baseline again after increase or decrease in blood glucose (Tbaseline) | 0-180 min
Total area under curve from 0 to 180 min for blood glucose concentration (AUC(0-180min)) | 0-180 min
Baseline corrected area under curve from 0 to 180 min for blood glucose concentration (AUCbase_c(0-180min)) | 0-180 min
  Area under curve from 0 to 180 min minus baseline*180min
Adverse events (AEs) | After screening till study day 22 (+24 hours)
Gastrointestinal tolerability (assessed by subject's questionnaire) | 180 min
Gastrointestinal tolerability (assessed by subject's questionnaire) | 24 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Menzel, MD, Principal Investigator — CRO BioTeSys GmbH
Locations (1):
- CRO BioTeSys GmbH, Esslingen am Neckar, Germany

IPD SHARING:
Plan to Share IPD: No